CLINICAL TRIAL: NCT02351739
Title: Randomized Phase 2 Trial of ACP-196 and Pembrolizumab Immunotherapy Dual CHECKpoint Inhibition In Platinum Resistant Metastatic Urothelial Carcinoma (RAPID CHECK Study)
Brief Title: Study of the Combination of ACP-196 and Pembrolizumab in Subjects With Platinum Resistant Urothelial Bladder Cancer
Acronym: KEYNOTE143
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-ST-005
Record Dates: First submitted 2015-01-28; First posted 2015-01-30 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pembrolizumab (Other): Arm 1: pembrolizumab monotherapy
  Interventions: Drug: pembrolizumab
- ACP-196 in combination with pembrolizumab (Other): Arm 2: ACP-196 in combination with pembrolizumab
  Interventions: Drug: ACP-196 in combination with pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab
  Arms: Pembrolizumab
Drug: ACP-196 in combination with pembrolizumab
  Arms: ACP-196 in combination with pembrolizumab

SUMMARY:
Study of the Combination of ACP-196 and Pembrolizumab in Subjects With Platinum Resistant Metastatic Urothelial Cancer

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Histologically or cytologically confirmed urothelial carcinoma of the bladder or mixed histology bladder cancer
* Metastatic bladder cancer with disease progression on or after platinum-based chemotherapy
* Any primary site of urothelial carcinoma including upper tract, renal pelvis, bladder, and ureters
* Prior therapy with ≥ 1 systemic chemotherapy regimens for urothelial carcinoma
* Presence of radiographically measurable disease (defined as the presence of ≥ 1 lesion that measures ≥ 10 mm [≥ 15 mm for lymph nodes]
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Prior malignancy (other than bladder cancer), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years of which will not limit survival to < 2 years.
* Known central nervous system metastases and/or carcinomatous meningitis
* Malabsorption syndrome, disease significantly affecting gastrointestinal function
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (7):
- United States (7):
  - University of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Durham, North Carolina
  - James Cancer Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Pembrolizumab Monotherapy: Arm 1: Pembrolizumab 200mg Administered as an intravenous (IV) infusion every 3 weeks (Q3W)
- Arm 2- Acalabrutinib+Pembrolizumab: Arm 2: Acalabrutinib 100mg PO BID plus Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W)
Period: Overall Study
Arm/Group | Arm 1: Pembrolizumab Monotherapy | Arm 2- Acalabrutinib+Pembrolizumab
Started | 38 | 40
Enrolled | 38 | 40
Received Study Medication | 35 | 40
Discontinued Study | 38 | 40
Completed | 0 | 0
Not Completed | 38 | 40

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab: Arm 1: pembrolizumab monotherapy
  pembrolizumab
- ACP-196 in Combination With Pembrolizumab: Arm 2: ACP-196 in combination with pembrolizumab
  ACP-196 in combination with pembrolizumab
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | ACP-196 in Combination With Pembrolizumab | Total
Number analyzed (Participants) | 35 | 40 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (11.08) | 66.4 (8.53) | 66.1 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 34 | 40 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 32 | 37 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Every 12 weeks for up to 2 years.
Population: The study participants had to have a minimum of one scan (for tumor assessment) after randomization/treatment in order to be considered analyzed.
  And some of the participants didn't make it to Wk 7 of treatment, hence reduction in the number of subjects analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | ACP-196 in Combination With Pembrolizumab
Number analyzed (Participants) | 31 | 34
Participants | 9 | 8

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after Day 0 and on or before Day 730.
Groups:
- Arm 1 - Pembrolizumab Monotherapy: Arm 1: Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W)
- Arm 2 - Acalabrutinib+Pembrolizumab: Arm 2: Acalabrutinib 100mg PO BID plus Pembrolizumab 200mg administered as an intravenous (IV) infusion every 3 weeks (Q3W)
Arm/Group | Arm 1 - Pembrolizumab Monotherapy | Arm 2 - Acalabrutinib+Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 25/35 | 31/40
Serious Adverse Events (participants affected / at risk) | 15/35 | 23/40
Other Adverse Events (participants affected / at risk) | 34/35 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Pembrolizumab Monotherapy (N=35) | Arm 2 - Acalabrutinib+Pembrolizumab (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Autoimmune Colitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1 — General Disorders and Administration Site Conditions
Pyrexia (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions
Pain (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions
Autoimmune Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Immune-Mediated Hepatitis (Hepatobiliary disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 3
Urinary Tract Infection (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Peritonitis Bacterial (Infections and infestations) | 1 | 0
Systemic Candida (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1
Radiation Proctitis (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Aspartate Aminotransferase (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute Kidney Disease (Renal and urinary disorders) | 2 | 5
Haematuria (Renal and urinary disorders) | 1 | 2
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Pembrolizumab Monotherapy (N=35) | Arm 2 - Acalabrutinib+Pembrolizumab (N=40)
Anaemia (Blood and lymphatic system disorders) | 8 | 13
Tachycardia (Cardiac disorders) | 1 | 4
Atrial Fibrillation (Cardiac disorders) | 0 | 2
Sinus Tachycardia (Cardiac disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 6 | 3
Vision Blurred (Eye disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 10 | 13
Diarrhea (Gastrointestinal disorders) | 7 | 16
Nausea (Gastrointestinal disorders) | 11 | 10
Constipation (Gastrointestinal disorders) | 5 | 12
Abdominal Pain (Gastrointestinal disorders) | 6 | 10
Abdominal Distension (Gastrointestinal disorders) | 4 | 3
Dry Mouth (Gastrointestinal disorders) | 3 | 3
Dysepsia (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 16 | 34 — General Disorders and Administration Site Conditions
Pyrexia (General disorders) | 6 | 10 — General Disorders and Administration Site Conditions
Oedema Peripheral (General disorders) | 4 | 7 — General Disorders and Administration Site Conditions
Chills (General disorders) | 2 | 3 — General Disorders and Administration Site Conditions
Non-Cardiac Chest pain (General disorders) | 1 | 4 — General Disorders and Administration Site Conditions
Asthenia (General disorders) | 2 | 2 — General Disorders and Administration Site Conditions
Gait Disturbance (General disorders) | 3 | 1 — General Disorders and Administration Site Conditions
Peripheral Swelling (General disorders) | 3 | 1 — General Disorders and Administration Site Conditions
Chest Pain (General disorders) | 1 | 2 — General Disorders and Administration Site Conditions
Urinary Tract Infection (Infections and infestations) | 9 | 7
Candida Infection (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 1
Rhinitis (Infections and infestations) | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 6 | 5
Contusion (Injury, poisoning and procedural complications) | 2 | 3
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 | 0
Alanine Aminotransferase Increased (Investigations) | 3 | 14
Aspartate Aminotransferase Increased (Investigations) | 2 | 11
Weight Decreased (Investigations) | 3 | 8
Blood Creatinine Increased (Investigations) | 5 | 5
Amylase Increased (Investigations) | 1 | 4
Lipase Increased (Investigations) | 1 | 4
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 4
Platelet Count Decreased (Investigations) | 0 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 14 | 16
Dehydration (Metabolism and nutrition disorders) | 1 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 4 | 8
Dizziness (Nervous system disorders) | 4 | 6
Dysgeusia (Nervous system disorders) | 1 | 4
Neuropathy Peripheral (Nervous system disorders) | 3 | 2
Paraesthesia (Nervous system disorders) | 2 | 2
Presyncope (Nervous system disorders) | 1 | 3
Balance Disorder (Nervous system disorders) | 0 | 2
Dizziness Postural (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 6 | 4
Insomnia (Psychiatric disorders) | 2 | 7
Confusional State (Psychiatric disorders) | 2 | 4
Depression (Psychiatric disorders) | 3 | 2
Haematuria (Renal and urinary disorders) | 2 | 4
Dysuria (Renal and urinary disorders) | 4 | 1
Acute Kidney Injury (Renal and urinary disorders) | 2 | 2
Bladder Spasm (Renal and urinary disorders) | 2 | 2
Urinary Retention (Renal and urinary disorders) | 2 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 5
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4 | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 3
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 2
Skin Discoloration (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2
Hypotension (Vascular disorders) | 6 | 8
Hypertension (Vascular disorders) | 2 | 3
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-05-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT02351739/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT02351739/SAP_001.pdf